CLINICAL TRIAL: NCT06967480
Title: MG-EVOLUTION. Early Ravulizumab Treatment Of Anti- AChR Antibody-Positive Generalized Myasthenia Gravis: A Real-World Study With Biomarker Analysis
Brief Title: Early Ravulizumab Treatment Of Anti- AChR Antibody-Positive Generalized Myasthenia Gravis
Status: Recruiting | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D9281R00002
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Generalized Myasthenia Gravis; Anti-AChR Antibody Positive
Keywords: Anti-AChR Antibody-Positive; Generalized Myasthenia Gravis; gMG; Ravulizumab
MeSH Terms: conditions — Myasthenia Gravis | interventions — ravulizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ravulizumab: Participants will receive Ravulizumab until Week 50 ± 14 days after baseline or until discontinuation.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — Participants will receive Ravulizumab.

SUMMARY:
The primary objective of the study is to evaluate the effectiveness of Ravulizumab in improving MG-ADL in an early-stage AChR+ gMG population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MG confirmed by:

  * History of a positive serologic test for anti-AChR antibodies, and
  * One of the following:

    * History of abnormal neuromuscular transmission test demonstrated by singlefibre electromyography or repetitive nerve stimulation
    * History of positive anticholinesterase test (e.g., edrophonium chloride test); or
    * Patient demonstrated improvement in MG signs on oral cholinesterase inhibitors, as assessed by the treating physician
* Disease duration from MG onset ≤ 3 years before T-4 (Enrolment);
* MGFA class IIb to IV;
* Patient eligible for Ravulizumab treatment based on AIFA reimbursement criteria
* Vaccination cycle for Neisseria meningitidis completed at least two weeks before Ravulizumab initiation or antibiotics chemoprophylaxis according to the SmPC.

Exclusion Criteria:

* Patient unable to understand and sign the informed consent
* Hypersensitivity to the active substance or to any of the excipients of the study product
* Patient for whom the study product is contraindicated according to SmPC
* Previous treatment with C5 inhibitors
* Last rituximab infusion performed < 6 months before T-4 (Enrolment)
* Last infusion with FcRn blockers performed < 3 months before T-4 (Enrollment)
* Pregnant or lactating or planning a pregnancy during the study
* Patient who plan to relocate during the study
* Patient who are unsure of following the visit schedule
* Patient unable to complete questionnaires
* Previous or current participation to other interventional studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anti-AChR antibody positive, generalized, myasthenia gravis elegible to Ravulizumab treatment with a disease duration from onset equal or less than 3 years.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Myasthenia Gravis-Activities of Daily Living (MG-ADL) Total Score at Week 50 | Week 50
Change From Baseline in MG-ADL Total Score at Week 50 | Baseline, Week 50

SECONDARY OUTCOMES:
MG-ADL Total Score at Weeks 2, 10, and 26 | Weeks 2, 10, and 26
Change From Baseline in MG-ADL Total Score at Weeks 2, 10 and 26 | Baseline, Weeks 2, 10 and 26
Percentage of Participants With >=2- Point Reduction From Baseline in MG-ADL Total Score at Weeks 2, 10, 26, and 50 | Baseline, Weeks 2, 10, 26, and 50
Quantitative Myasthenia Gravis (QMG) Total Score at Weeks 2, 10, 26, and 50 | Weeks 2, 10, 26, and 50
Change From Baseline in QMG Total Score at Weeks 2, 10, 26 and 50 | Baseline, Weeks 2, 10, 26 and 50
Percentage of Participants With >=3- Point Reduction From Baseline in QMG Total Score at Weeks 2, 10, 26, and 50 | Baseline, Weeks 2, 10, 26, and 50
Myasthenia Gravis Composite (MGC) Total Score at Weeks 2, 10, 26, and 50 | Weeks 2, 10, 26, and 50
Change From Baseline in MGC Total Score at Weeks 2,10, 26 and 50 | Baseline, Weeks 2, 10, 26 and 50
Percentage of Participants With >=3- Point Reduction From Baseline in MGC Total Score at Weeks 2, 10, 26 and 50 | Baseline, Weeks 2, 10, 26, and 50
Myasthenia Gravis Quality of Life 15-Item Scale - Revised (MG-QoL15r) Total Score at Weeks 10, 26, and 50 | Weeks 10, 26, and 50
Change From Baseline in MG-QoL15r Total Score at Weeks 10, 26 and 50 | Baseline, Weeks 10, 26 and 50
Hospital Anxiety and Depression Scale (HADS) Total Score at Weeks 10, 26, and 50 | Weeks 10, 26, and 50
Change From Baseline in HADS Total Score at Weeks 10, 26 and 50 | Baseline, Weeks 10, 26 and 50
Insomnia Severity Index Scale (ISI) Total Score at Weeks 10, 26, and 50 | Weeks 10, 26, and 50
Change From Baseline in ISI Total Score at Weeks 10, 26 and 50 | Baseline, Weeks 10, 26 and 50
Pain Visual Analogue Scale (Pain VAS) Total Score at Weeks 2, 10, 26, and 50 | Weeks 2, 10, 26, and 50
Change From Baseline in Pain VAS Total Score at Weeks 2, 10, 26 and 50 | Baseline, Weeks 2, 10, 26 and 50
Percentage of Participants With Mean Dose Reduction From Baseline of Corticosteroids and Immunosuppressants (ISTs) Treatment at Weeks 2, 10, 26, and 50 | Baseline, Weeks 2, 10, 26, and 50
Percentage of Participants in Different ISTs Status at Baseline, and at Weeks 2, 10, 26, and 50 | Baseline, Weeks 2, 10, 26, and 50
Number of Clinical Deterioration Events | Baseline, Weeks 2, 10, 26, and 50
Percentage of Participants With Minimal Symptom Expression at Weeks 2, 10, 26, and 50 | Weeks 2, 10, 26, and 50
Institute For Medical Technology Assessment (iMTA) Productivity Cost Questionnaire (iPCQ) Score at Weeks 10, 26, and 50 | Weeks 10, 26, and 50
Change From Baseline in iMTA iPCQ Score at Weeks 10, 26 and 50 | Baseline, Weeks 10, 26 and 50
Biomarkers analyses (complement system proteins, interleukins and miRNA serum levels) | Baseline, Week 10, 26, and 50

CONTACTS AND LOCATIONS:
Locations (21):
- Italy (21):
  - Clinical Trial Site, Bergamo
  - Clinical Trial Site, Bologna
  - Clinical Trial Site, Brescia
  - Clinical Trial Site, Florence
  - Clinical Trial Site, Imperia
  - Clinical Trial Site, Lecco
  - Clinical Trial Site, Messina
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Napoli
  - Clinical Trial Site, Novara
  - Clinical Trial Site, Orbassano
  - Clinical Trial Site, Padua
  - Clinical Trial Site, Palermo
  - Clinical Trial Site, Parma
  - Clinical Trial Site, Pavia
  - Clinical Trial Site, Pisa
  - Clinical Trial Site, Roma
  - Clinical Trial Site, Salerno
  - Clinical Trial Site, San Giovanni Rotondo
  - Clinical Trial Site, Sassari
  - Clinical Trial Site, Torino

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR